CLINICAL TRIAL: NCT05881707
Title: A Randomized, Open-label, Single Dose, 4-period Replicate Crossover Study to Evaluate the Pharmacokinetic Profiles and Safety of CKD-828 in Healthy Volunteers Under Fasting Conditions
Brief Title: A Clinical Trial to Compare the Pharmacokinetic and Safety of CKD-828 20/1.25mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A30_18BE2304
Record Dates: First submitted 2023-05-21; First posted 2023-05-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — 2-(3,4-dimethoxyphenyl)-8-(4-hydroxy-3-methoxyphenyl)-6-methyl-2-isopropyl-6-azaoctanitrile

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): * Period 1: D064, D702 - A single oral dose of 2 tablets
  * Period 2: CKD-828 - A single oral dose of 1 tablet
  * Period 3: D064, D702 - A single oral dose of 2 tablets
  * Period 4: CKD-828 - A single oral dose of 1 tablet
  Interventions: Drug: CKD-828, D064, D702
- Sequence 2 (Experimental): * Period 1: CKD-828 - A single oral dose of 1 tablet
  * Period 2: D064, D702 - A single oral dose of 2 tablets
  * Period 3: CKD-828 - A single oral dose of 1 tablet
  * Period 4: D064, D702 - A single oral dose of 2 tablets
  Interventions: Drug: CKD-828, D064, D702

INTERVENTIONS:
Drug: CKD-828, D064, D702 — QD, PO

SUMMARY:
A clinical trial to compare the pharmacokinetic and safety of CKD-828 20/1.25mg

DETAILED DESCRIPTION:
A randomized, open-label, single dose, 4-period replicate crossover study to evaluate the pharmacokinetic profiles and safety of CKD-828 in healthy volunteers under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult aged ≥ 19 and <55 at screening
2. Those who have a body mass index (BMI) of not less than 18.0 kg/m2 and not more than 30.5 kg/m2 and weigh not less than 55 kg
3. A person who has no congenital or chronic disease within the last three years and has no pathological symptoms or findings as a result of medical examination
4. A person who is deemed suitable for testing as a result of laboratory tests (hematological tests, hemochemistry tests, urinary tests, virus/bacterial tests, etc.) conducted by the tester according to the characteristics of the drug, vital signs, electrocardiogram tests, etc
5. A person who has signed a written consent approved by the Chonbuk National University Hospital Clinical Trial Review Board (IRB) after fully explaining the purpose, contents, etc. of the test before participating in the test
6. A person who has agreed not to donate sperm during the pre-clinical period and one month after taking the last clinical drug (non-hormonal contraceptive method: condom use, intrauterine device (IUD, IUS), tubular ligation, cervical cap, contraceptive diaphragm, etc.)
7. A person who has the ability and will to participate during the pre-test period

Exclusion Criteria:

1. Clinically significant blood, kidneys (severe renal dysfunction, etc.), endocrine, respiratory, gastrointestinal, urology, cardiovascular (within one month of severe aortic stenosis, instability, or myocardial infarction), liver (severe hepatic dysfunction, biliary obstruction, bile congestion, etc.), mental, nerve or immune disease simple dental evidence
2. A person who has a history of gastrointestinal diseases (e.g., esophageal diseases such as esophageal dysphagia or esophageal stenosis, Crohn's disease) or surgery (excluding simple appendectomy, hernia, or extraction surgery) that can affect drug absorption
3. A person who shows the following figures as a result of performing an inspection laboratory inspection during screening

   * ALT or AST > Twice the upper limit of the normal range
   * CK> 3 times the upper limit of the normal range
   * eGFR <60 mL/min/1.73 m2 using CKD-EPI formula
4. Screening Those with a history of regular alcohol consumption exceeding 210 g/week within 6 months (Beer (5%) 1 glass (250 mL) = 10 g, Soju (20%) 1 glass (50 mL) = 8 g, Wine (12%) 1 glass (125 mL) = 12 g)
5. Smokers with 20 or more cigarettes per day within 6 months of screening
6. A person who has taken another clinical trial drug or biological equivalence test drug within six months prior to the first administration of the clinical trial drug
7. Person who falls under the following results of vital signs measurement during screening

   ☞ Those with systolic blood pressure of less than 90 mmHg, 140 mmHg or more, or diastolic blood pressure of less than 60 mmHg or 90 mmHg or more in the sedentary state
8. A person who has a history of serious alcohol or drug misuse within one year of screening
9. A person who has taken a drug known to significantly induce or inhibit drug metabolites within 30 days prior to the first administration of a drug for clinical trials
10. A person who has taken prescription or non-prescription drugs within 10 days prior to the first administration of a clinical trial drug
11. A person who has donated all blood within two months before the first administration of a clinical trial drug, or has donated blood components within one month, or received a blood transfusion within one month
12. Those with severe acute/chronic medical and mental conditions that may increase risk or interfere with the interpretation of test results due to the administration and participation in clinical trial drugs
13. A person who has overreaction to clinical trial drugs, the main ingredients and components of clinical trial drugs, or other dihydropyridine-based drugs
14. Patients with hereditary angioedema or patients with a history of angioedema when treated with ACE inhibitors or angiotensin II receptor antagonists
15. Shock patients (including cardiac shock)
16. Pregnant or lactating women
17. Other persons deemed inappropriate by the tester to participate in this test

Ages: 19 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-07-04 (Actual); Primary Completion 2023-09-02 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
AUCt of CKD-828 | Pre-dose(0 hour), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Area under the concentration-time curve time zero to time
Cmax of CKD-828 | Pre-dose(0 hour), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Maximum plasma concentration of the drug

CONTACTS AND LOCATIONS:
Overall Officials: Mingul Kim, Ph.D, Principal Investigator — Jeonbuk National University Hospital
Locations (1):
- Jeonbuk National University Hospital, Seoul, South Korea